CLINICAL TRIAL: NCT03554564
Title: Project VOICE: Vascular Outcomes Improvement Through Collection of PatiEnt Reported Data
Acronym: VOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wake Forest University (Other); Vascular Cures (Other)
Responsible Party: Principal Investigator, Matthew Corriere, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00142561; HUM00142561 (Other: University of Michigan IRB)
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; claudication; supervised exercise therapy; walking; quality of life
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Voice

STUDY DESIGN:
Intervention Model Description: Randomized, non-blinded crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOICE/Fitbit (Experimental): VOICE enrollment with Fitbit walking activity tracking. During the VOICE phase, participants will use the digital health platform that integrates PAD-specific educational content, surveys, and Fitbit walking activity tracking for a total of five weeks (one week run-in phase plus four week study phase).
  Interventions: Behavioral: VOICE/Fitbit
- Daily self-reported exercise adherence (Other): Usual care prescribed by physician (walking exercise instructions). During the Usual Care control phase, participants will conduct walking exercise based on instructions received in clinic. Walking exercise will be tracked and self-reported by participants, using a written calendar log. Participants will not have access to the VOICE platform, or use of Fitbit technology during this phase.
  Interventions: Other: Daily self-reported exercise adherence

INTERVENTIONS:
Behavioral: VOICE/Fitbit — During the VOICE (intervention) phase, participants will use the digital health platform plus Fitbit walking activity tracking for a total of five weeks (one week run-in phase plus four week study phase)
  Other Names: Digital health platform plus tracked exercise
  Arms: VOICE/Fitbit
Other: Daily self-reported exercise adherence — During usual care, patients will self-report on a daily basis if they met the walking exercise goal consistent with instructions from their clinician. Self-report will be recorded as a daily categorical (yes/no) variable.
  Arms: Daily self-reported exercise adherence

SUMMARY:
The purpose of this study is to evaluate the feasibility of a digital health platform coupled with walking activity tracking for patients with Peripheral Artery Disease (PAD) and symptoms limited to claudication.

DETAILED DESCRIPTION:
This is a two center, non-blinded, 2 period randomized crossover trial. 50 patient subjects are planned. Patient participants will be identified and recruited from clinical environments (including clinics and diagnostic testing departments) at participating sites. Diagnosis and testing will occur through usual clinical care, and participants will not incur financial costs related to participation. A crossover design will be utilized, where all participants will use the VOICE platform with activity tracking for 35 days and usual care for 30 days. Randomization will determine the order in which participation in the VOICE phase versus the usual care phase occur. Randomization will occur using a closed envelope system. For patients in the VOICE platform group, data collection will occur over a total of 35 days, including an initial 5-day "run in" period during which participants will orient themselves to the system. Each provider participant will receive a single end-user survey evaluating VOICE from their perspective.

Screening of patients electronic medical records will be done to determine subject eligibility. Subjects who meet all inclusion criteria will be approached to participate.

Total duration of subject participation will be 9 weeks during the control and intervention phases, with a final follow-up survey at 6 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic PAD with claudication
* Ankle- brachial index (ABI) ≤ 0.9 or non-compressible leg arteries
* Walking exercise therapy recommended as treatment for PAD by the healthcare provider
* Willingness to be randomized to VOICE platform or control group
* Ability to access the internet
* Willing to sign an informed consent

Exclusion Criteria:

* Walking exercise therapy not recommended due to contraindication or any other reason
* Wheelchair dependence or inability to walk unassisted
* Presence of foot ulcers, wounds, or gangrene
* History of major extremity amputation
* Lack of objective physiologic data validating PAD diagnosis
* Claudication symptoms due to diagnoses other than PAD (i.e., popliteal entrapment syndrome)
* Inability to speak or read English
* Severe mental illness
* Inability to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Walking adherence (days with walking exercise/total days per study period) | 2 months
  Self-reported walking adherence based on a daily log will be compared with exercise assessed using tracked walking activity during the VOICE/Fitbit phase. Adherence will be evaluated based on number of days during the study period where walking exercise was performed, and will be evaluated as a categorical (yes/no) variable.

SECONDARY OUTCOMES:
Tracked Walking Activity: Distance (meters) | 2 months
  Distance in kilometers/miles recorded by Fitbit during VOICE intervention phase.
Tracked Walking Activity: Steps (count) | 2 months
  Number of steps recorded by Fitbit device during VOICE intervention phase.
Tracked Walking Activity: Time (minutes) | 2 months
  Number of minutes/hours recorded by Fitbit during VOICE intervention phase.
Tracked Walking Activity: Cadence (steps per minute) | 2 months
  Average steps per minute recorded by Fitbit during VOICE intervention phase.
Sleep interruption (mean nightly frequency) | 2 months
  While in VOICE/Fitbit phase, user data is collected by the unit for each sleep cycle including sleep duration, schedule, and quality. The data collected also shows insight into the number of sleep disruptions, restless periods, and minutes awake. This will only be tracked and recorded using Fitbit for the duration of the VOICE/Fitbit intervention phase.
PROMIS Pain Interference Short Form 6a (raw score, T-score conversion) | 1 month, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System designed to gauge the level to which pain interferes with the participant's social, work, and day-to-day household activities. This six-item assessment yields total values ranging from 4 (low) to 20 (high) based on reported severity of pain interference, within a seven day duration. This measure will be repeated three times across the study and the data will be analyzed to determine consistency, improvement, and/or deterioration of quality.
PROMIS Physical Function Short Form 6b (raw score, T-score conversion) | 1 month, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System short form questionnaire designed to gauge the level to which the participant feels their disease limits their ability to perform daily tasks and activities, at the time of the assessment. This six-item questionnaire yields total values ranging from 6 to 30, with a higher score representing a higher level of functional ability. This measure will be repeated three times across the study and the data will be analyzed to determine consistency, improvement, and/or deterioration of quality.
PROMIS Sleep Disturbance Short Form 4a (raw score, T-score conversion) | 1 month, 2 months, 6 months
  Patient-Reported Outcomes Measurement Information System is a short form questionnaire administered to participants to gauge sleep depth and quality, within a seven day duration. This nine-item assessment is a combination of items in which participants are asked to respond either affirmatively or negatively, and with a subset of questions scored on a numerical scale with a raw score ranging from 4 (low) to 20 (high). This measure will be repeated three times across the study and the data will be analyzed to determine consistency, improvement, and/or deterioration of quality.
VascuQol-6 | 1 month, 2 months, 6 months
  The Vascular Quality of Life Questionnaire, or VascuQoL-6, is a disease-specific instrument in which the participant is asked about their concerns, abilities, and activities, referencing the previous two-week time frame. Overall values can range from 6 to 24 for the VascuQoL-6, with a higher total sum representing better participant health. This measure will be repeated three times across the study and the data will be analyzed to determine consistency, improvement, and/or deterioration of quality.

OTHER OUTCOMES:
Grip Strength (kg) | Baseline
  Dominant hand grip strength will be measured and recorded by study staff, using a Jamar hand dynamometer. The participant will be directed to squeeze the unit's handle to obtain a "peak-hold" reading, with a potential isometric grip force ranging from 0-200lbs (90kgs). The numerical output will be recorded as part of the participant's chart to be analyzed and compared with the investigator's data set.
Ankle-Brachial Index | Baseline
  Ankle-brachial index (ABI) is a diagnostic measure used by providers to determine the likelihood and severity of blocked arteries, due to peripheral artery disease. ABI is calculated by comparing the ratio of the recorded blood pressure at a participant's ankle to the pressure in the upper arm. Participant's previous ABI values in MiChart will be used to determine eligibility at time of enrollment. Newly ordered ABI studies will then be tracked by study staff and recorded to be analyzed with the data set, for the duration of their participation in the study.
Diagnostic Tests | 6 months
  PAD-specific imaging or diagnostic tests (based on electronic medical record)
PAD treatment interventions | 6 months
  Any clinical treatment interventions performed during the study period will be captured, including: initiation of symptomatic pharmacotherapy, procedures related to PAD (including lower extremity CTA, MRA, angiography, revascularization procedures, or surgical procedures). This outcome will be assessed using the patient electronic medical record in addition to patient self-report.
Walking goal (steps per day) | baseline
  Steps per day selected as walking goal at initiation of the VOICE/Fitbit phase
Change in walking goal (steps per day) | 2 months
  At completion of the VOICE/Fitbit phase, participants will be asked if they changed their daily walking goal from baseline. The updated (new) goals will be recorded for those who respond "yes".

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A. Corriere, M.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan - Vascular Surgery Section, Ann Arbor, Michigan
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided